CLINICAL TRIAL: NCT00870363
Title: A Pilot Project of Virologic, Pharmacologic and Immunologic Correlates of Gastrointestinal-Associated Lymphoid Tissue Immune Reconstitution Following Maraviroc Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200816535
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections
Keywords: HIV; HIV positive; Gastrointestinal Associated Lymphoid Tissue (GALT); GALT Immune Reconstruction; treatment naive
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — Maraviroc; Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): maraviroc in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Interventions: Drug: maraviroc in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor)
- 2 (Active Comparator): maraviroc PLUS raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Interventions: Drug: maraviroc plus raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor)
- 3 (Active Comparator): efavirenz or other NNRTI (non-nucleoside reverse transcriptase inhibitor) in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Interventions: Drug: efavirenz [or other NNRTI (non-nucleoside reverse transcriptase inhibitor)]
- 4 (No Intervention): HIV-negative

INTERVENTIONS:
Drug: maraviroc in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) — maraviroc 300mg 1 tablet taken twice a day without regard to food taken in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Other Names: Selzentry
  Arms: 1
Drug: maraviroc plus raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) — maraviroc 300mg 1 tablet taken twice a day without regard to food PLUS raltegravir 400mg 1 tablet taken twice a day without regard to food in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Other Names: Selzentry (maraviroc)
  Arms: 2
Drug: efavirenz [or other NNRTI (non-nucleoside reverse transcriptase inhibitor)] — efavirenz 600mg 1 capsule is taken once a day without regard to food in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  Other Names: Sustiva
  Arms: 3

SUMMARY:
This research study is being done to find out how the immune system in the small intestines improves after taking antiretroviral (anti-HIV) medications. Biopsies (small snips of tissue) will be taken from the part of the intestines just below the stomach, and will be studied in the laboratory. The main purpose of this study is to measure the increase in the numbers of immune cells in the intestines to see if this number is related to the amount of medication that reaches the intestinal tissue, and the amount of virus that is still hiding there.

Subjects are either normal control subjects without HIV or, are HIV positive and are about to start HIV medications. As part of this study, HIV positive patients will be randomized to receive one of three possible combinations of medications.

1. maraviroc (Selzentry) in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) or
2. maraviroc PLUS raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) or
3. efavirenz (Sustiva) in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor)

Both Maraviroc and Raltegravir each represent new classes of medications in the way that they interfere with HIV making copies of itself. Maraviroc attaches to the surface of the T-cell that the virus uses to get into the cell and is therefore known as an entry inhibitor. Raltegravir blocks the virus from inserting itself into the DNA of the infected cell's nucleus and is therefore known as an Integrase Inhibitor. We hope to learn more about how antiretroviral drugs affect T cells and how immune function restores itself when HIV infection is treated.

DETAILED DESCRIPTION:
Despite improved survival, durable virologic suppression, and increases in peripheral CD4+ T-cell counts in patients receiving potent antiretroviral therapy (ART), immune reconstitution remains incomplete as measured by a number of additional surrogate markers. Perhaps critically important among areas of apparent incomplete immune recovery is the gastrointestinal-associated lymphoid tissue (GALT), where CD4+ T-cells repopulate very slowly if at all. Several new classes of antiretrovirals (ART) have recently been approved by the FDA that offer potential advantages in terms of immune reconstitution and/or the kinetics viral suppression over traditionally available treatment regimens. Maraviroc is a new ART agent from a novel class of HIV inhibitors, entry inhibitors, that results in rapid suppression of HIV and recovery of peripheral CD4+ T-cells. This project proposes to examine whether volunteers receiving maraviroc recover GALT immune cells more completely that those taking comparator ART. Raltegravir is an integrase inhibitor that blocks incorporation of the proviral HIV DNA into the host chromosomes leading to more rapid declines in plasma HIV load than has previously been observed. This project proposes to examine whether volunteers receiving maraviroc or maraviroc plus raltegravir recover GALT immune cells more completely that those taking comparator ART. An additional attraction of the use of maraviroc and raltegravir together is that they may provide a potent combination that is also lipid neutral and thereby constitute a 'Heart friendly HAART' (Highly Active Antiretroviral Therapy).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 18 years to 60 years inclusive
* HIV positive (no anticipated antiretroviral therapy adjustments/changes)
* CD4 count greater than or equal to 50 cells/ml within 30 days of screening
* CCR5 tropism by Trofile ES(TM)
* Can be on secondary prophylaxis with a history of AIDS defining illness
* All females of child-bearing potential must agree to use barrier methods to prevent pregnancy or be abstinent from sexual activity while on study.
* willing to sign consent form
* HIV Negative individuals will also be recruited for this study as a Control Group

Exclusion Criteria:

* allergy to peanuts or soya (maraviroc contains soya lecithin)
* abnormal coagulation parameters (PT greater than or equal to 1.2 ULN)
* thrombocytopenia (platelet count less than 50,000 within 6 weeks)
* known GI pathology
* contra-indications to upper endoscopy or conscious sedation
* anemia greater than grade 1
* any active acute opportunistic infection (OI) or therapy for acute OI within 30 days of entry into study
* positive pregnancy test
* aspirin, ibuprofen, warfarin, or other agents that interfere with the coagulation cascade taken within 1 week of endoscopy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Asmuth, MD, Principal Investigator — University of California, Davis Health System
Locations (1):
- CARES Clinic, Sacramento, California, United States

REFERENCES:
- [Result] Serrano-Villar S, Sainz T, Ma ZM, Utay NS, Chun TW, Mann S, Kashuba AD, Siewe B, Albanese A, Troia-Cancio P, Sinclair E, Somasunderam A, Yotter T, Deeks SG, Landay A, Pollard RB, Miller CJ, Moreno S, Asmuth DM. Correction: Effects of Combined CCR5/Integrase Inhibitors-Based Regimen on Mucosal Immunity in HIV-Infected Patients Naive to Antiretroviral Therapy: A Pilot Randomized Trial. PLoS Pathog. 2016 Mar 25;12(3):e1005540. doi: 10.1371/journal.ppat.1005540. eCollection 2016 Mar. No abstract available. PMID 27015639
- [Derived] Serrano-Villar S, de Lagarde M, Vazquez-Castellanos J, Vallejo A, Bernadino JI, Madrid N, Matarranz M, Diaz-Santiago A, Gutierrez C, Cabello A, Villar-Garcia J, Blanco JR, Bisbal O, Sainz T, Moya A, Moreno S, Gosalbes MJ, Estrada V. Effects of Immunonutrition in Advanced Human Immunodeficiency Virus Disease: A Randomized Placebo-controlled Clinical Trial (Promaltia Study). Clin Infect Dis. 2019 Jan 1;68(1):120-130. doi: 10.1093/cid/ciy414. PMID 29788075
- [Derived] Asmuth DM, Thompson CG, Chun TW, Ma ZM, Mann S, Sainz T, Serrano-Villar S, Utay NS, Garcia JC, Troia-Cancio P, Pollard RB, Miller CJ, Landay A, Kashuba AD. Tissue Pharmacologic and Virologic Determinants of Duodenal and Rectal Gastrointestinal-Associated Lymphoid Tissue Immune Reconstitution in HIV-Infected Patients Initiating Antiretroviral Therapy. J Infect Dis. 2017 Oct 17;216(7):813-818. doi: 10.1093/infdis/jix418. PMID 28968888
- [Derived] Ellis CL, Ma ZM, Mann SK, Li CS, Wu J, Knight TH, Yotter T, Hayes TL, Maniar AH, Troia-Cancio PV, Overman HA, Torok NJ, Albanese A, Rutledge JC, Miller CJ, Pollard RB, Asmuth DM. Molecular characterization of stool microbiota in HIV-infected subjects by panbacterial and order-level 16S ribosomal DNA (rDNA) quantification and correlations with immune activation. J Acquir Immune Defic Syndr. 2011 Aug 15;57(5):363-70. doi: 10.1097/QAI.0b013e31821a603c. PMID 21436711

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc in Combination With 2 NRTIs: maraviroc in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  maraviroc in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor): maraviroc 300mg 1 tablet taken twice a day without regard to food taken in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
- Maraviroc PLUS Raltegravir in Combination With 2 NRTIs: maraviroc PLUS raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  maraviroc plus raltegravir in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor): maraviroc 300mg 1 tablet taken twice a day without regard to food PLUS raltegravir 400mg 1 tablet taken twice a day without regard to food in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
- Efavirenz or Other NNRTI With 2 NRTIs: efavirenz or other NNRTI (non-nucleoside reverse transcriptase inhibitor) in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
  efavirenz [or other NNRTI (non-nucleoside reverse transcriptase inhibitor)]: efavirenz 600mg 1 capsule is taken once a day without regard to food in combination with 2 NRTIs (dual nucleoside reverse transcriptase inhibitor) pre-determined with primary care physician
- HIV Negative Controls Not on ART: HIV-negative
Period: Overall Study
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Started | 10 | 11 | 11 | 12
Completed | 10 | 8 | 8 | 12
Not Completed | 0 | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART | Total
Number analyzed (Participants) | 10 | 8 | 8 | 12 | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [25 to 43] | 35 [27 to 40] | 37 [25 to 46] | 35 [29 to 42] | 37 [25 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 5 | 9
  Male | 7 | 7 | 8 | 7 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 5 | 4 | 1 | 1 | 11
  White | 5 | 3 | 5 | 9 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 8 | 12 | 38
CD4 T-Cell count [Median (Inter-Quartile Range); unit: CELLS/MM^3] | 441 [369 to 511] | 453 [334 to 713] | 322 [233 to 536] | NA [NA to NA] — not measured in the negative control cohort | 436 [283 to 572]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Density of CD3+/CD4+ Cells Per Cubic Millimeter at the Effector Sites in the Duodenal Tissues Following Antiretroviral Therapy Regimen
Description: immunohistochemistry for CD3+/CD4+ cells counted manually within the lamina propria
Time Frame: Baseline and nine months for 3 treatment cohorts and Baseline for the control group, which was only assessed at one time point
Population: numbers represent an increase from baseline for the 3 treatment cohorts and represent the absolute value for the control group who were only measured at one timepjoint.
Measure: Mean (95% Confidence Interval); unit: cells/mm^2
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 10 | 8 | 8 | 12
cells/mm^2 | 24 [-44 to 92] | 89 [51 to 127] | 119 [-7 to 245] | 566 [509 to 688]
Statistical Analysis 1: Comparison: Maraviroc in Combination With 2 NRTIs vs Maraviroc PLUS Raltegravir in Combination With 2 NRTIs vs Efavirenz or Other NNRTI With 2 NRTIs vs HIV Negative Controls Not on ART; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis

2. Secondary Outcome: Trough Plasma and Tissue Drug Levels in Volunteers at the Time of the Upper Endoscopy
Description: The reported drug level is for the primary ART agent for that cohort. For the maraviroc arm, maraviroc plasma and tissue levels are reported. For the maraviroc plus raltegravir arm, the raltegravir plasma and tissue levels are reported. For the efavirenz arm, the efavirenz plasma and tissue levels are reported. HIV negative controls were not on ART and did not have drug levels measured.
Time Frame: nine months
Population: HIV negative controls were not on ART and did not have drug levels measured.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 10 | 8 | 8 | 0
ng/mL
  plasma primary ART | 94.5 [60.5 to 126.5] | 397 [93.4 to 1131.3] | 2459 [1485.7 to 5328.2] |
  duodenal tissue primary ART | 0.7 [0.3 to 1.4] | 0.1 [0.07 to 0.3] | 11.1 [8.4 to 15.0] |

3. Secondary Outcome: Change in HIV DNA Per 10^6 Cells in Duodenal Tissue Versus PBMC by Drug Regimen Received
Description: single-cell suspension of digested duodenal tissue and Ficol-Hypaque separated PBMC underwent HIV-DNA PCR
Time Frame: Baseline and nine months
Population: HIV negative controls did not have HIV-DNA in blood or tissue
Measure: Mean (95% Confidence Interval); unit: copies/10^6 cells
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 10 | 8 | 8 | 0
copies/10^6 cells
  PBMC HIV-DNA | -1709 [-2845 to -573] | -2500 [-4868 to -132] | -1330 [-5354 to 2693] |
  Duodenal HIV-DNA | -16 [-40 to 8] | -846 [-1721 to 30] | -325 [-701 to 51] |

4. Secondary Outcome: Change in GALT CD4+ and CD8+ T-cell Subpopulations (naïve and Memory Subsets)
Time Frame: nine months
Population: data were not collected due to the samples not being suitable for the epitopes being measured
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Lymphocyte Immune Function and Activation at Two Time Points Approximately Nine Months Apart in GALT; and Four Timepoints (Month 0, 3, 6, and 9) in Peripheral Blood
Time Frame: nine months
Population: data were not collected due to inadequate sample volume for this complex experiment design
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Changes in CD4+ T-cell Numbers by Treatment Regimen
Description: peripheral absolute CD4+ T-cell counts increase from baseline to 9 months of cART by commercial assay
Time Frame: Baseline and nine months
Population: peripheral CD4 T-cell counts were not measured in the HIV negative cohort
Measure: Mean (95% Confidence Interval); unit: cells/mL
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 10 | 8 | 8 | 0
cells/mL | 221 [149 to 293] | 231 [134 to 327] | 194 [57 to 330] |

7. Secondary Outcome: Immune Reconstitution With Respect to Absolute Numbers of CD4+ T-cells, the Relative Proportion of T-cell Subpopulations in the Tissue, and Immune Activation to a Cohort of Normal Controls
Time Frame: nine months
Population: data was not collected/analyzed due to complications in the assays for immune activation in the collected samples
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: during the 9 months of the study participation
Arm/Group | Maraviroc in Combination With 2 NRTIs | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs | Efavirenz or Other NNRTI With 2 NRTIs | HIV Negative Controls Not on ART
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 1/11 | 1/11 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc in Combination With 2 NRTIs (N=10) | Maraviroc PLUS Raltegravir in Combination With 2 NRTIs (N=11) | Efavirenz or Other NNRTI With 2 NRTIs (N=11) | HIV Negative Controls Not on ART (N=12)
gastrointestinal intolerance (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — nausea due to medication that resolved with treatment modification
neuropsychiatric side effect (Nervous system disorders) | 0 | 0 | 1 | 0 — vivid dreams

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes